CLINICAL TRIAL: NCT00505284
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Trial to Evaluate the Efficacy and Safety of E2007 in Patients With Painful Diabetic Neuropathy
Brief Title: An Evaluation of the Efficacy and Safety of E2007 in Patients With Painful Diabetic Neuropathy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: Eisai Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E2007-G000-227; 2006-006488-22 (EudraCT Number)
Record Dates: First submitted 2007-07-20; First posted 2007-07-23 (Estimated); Results first posted 2013-02-08 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2013-02

CONDITIONS: Diabetic Neuropathy
Keywords: Diabetic neuropathy
MeSH Terms: conditions — Diabetic Neuropathies | interventions — perampanel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Perampanel 2mg (Active Comparator)
  Interventions: Drug: E2007 (2 mg)
- Perampanel 4mg (Active Comparator)
  Interventions: Drug: E2007 (4 mg)
- Perampanel 6mg (Active Comparator)
  Interventions: Drug: E2007 (6 mg)
- Perampanel 8mg (Active Comparator)
  Interventions: Drug: E2007 (8 mg)

INTERVENTIONS:
Drug: Placebo — Placebo tablets, once daily, for 15 weeks (taken orally).
  Arms: Placebo
Drug: E2007 (2 mg) — Perampanel, 2 mg once daily, for 15 weeks (taken orally).
  Other Names: Perampanel
  Arms: Perampanel 2mg
Drug: E2007 (4 mg) — Perampanel, 2 mg once daily for three weeks, followed by 4 mg, once daily, for 12 weeks (taken orally).
  Other Names: Perampanel
  Arms: Perampanel 4mg
Drug: E2007 (6 mg) — Perampanel, 2 mg once daily for three weeks, followed by 4 mg once daily, for three weeks and 6 mg, once daily, for nine weeks (taken orally).
  Other Names: Perampanel
  Arms: Perampanel 6mg
Drug: E2007 (8 mg) — Perampanel, 2 mg once daily, for three weeks, followed by 4 mg, once daily for three weeks, 6 mg once daily for three weeks and 8 mg, once daily, for six weeks (taken orally).
  Other Names: Perampanel
  Arms: Perampanel 8mg

SUMMARY:
The purpose of this study is to determine the efficacy and safety of Perampanel in patients with painful diabetic neuropathy.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, parallel-group study. This is a 5-arm, 21-week study comprised of up to a 2-week Screening period, a 15-week Dose-Escalation and Maintenance Phase using 4 doses of E2007 (2 mg, 4 mg, 6 mg, and 8 mg) or placebo, and a 4-week, single-blind placebo Follow-Up Phase. Patients will be randomly assigned to one of the five treatment groups. Those patients assigned to receive either 4 mg, 6 mg, or 8 mg E2007 will be escalated to the appropriate dose according to an escalation schedule. All patients will take four identical-looking tablets on a daily basis for the entire study duration for blinding purposes.

ELIGIBILITY:
INCLUSION CRITERIA:

To be included, patients must meet all of the following:

1. Provide written informed consent, prior to entering the study or undergoing any study procedures
2. Male and female patients ≥18 years of age will be eligible for enrollment. Females should be either not of childbearing potential as a result of surgery or menopause (1 year after onset), or of childbearing potential and practicing a medically acceptable method of contraception (e.g., abstinence, a barrier method plus spermicide, or intrauterine device [IUD]) for at least 1 month before Screening (Visit 1) and for 1 month after the end of the study (Visit 8). They must also have a negative serum beta-human chorionic gonadotropin (ß-hCG) at Screening (Visit 1). Those females using hormonal contraceptives must also be using an additional approved method of contraception (e.g., a barrier method plus spermicide or IUD) starting with the Baseline Phase and continuing throughout the study period.
3. Have Type I or Type II diabetes with painful, distal, symmetrical, sensory-motor neuropathy attributed to diabetes, of at least 12 months duration
4. Have pain that has been stable over the past 6 months and, in the opinion of the investigator, not in an identifiably improving or worsening trend
5. Have hemoglobin A1c ≤ 11%
6. Score of ≥ 40 mm on the visual analog scale (VAS) of the short form McGill Pain Questionnaire (SF-MPQ) at both Screening (Visit 1) and Baseline (Visit 2 prior to randomization)
7. Have completed the patient diary for at least 6 of the 7 days prior to Baseline (Visit 2)
8. Have average daily pain score of ≥ 4, on 11-point Likert-type numeric rating scale during the 7 days prior to Baseline (to be obtained from the patient diary)
9. Be reliable, willing, and able to cooperate with all study procedures including the following:

   1. accurately fill out the diary on a daily basis
   2. return for study visits on the required dates
   3. accurately and reliably report symptoms (including treatment-emergent signs and symptoms)
   4. take study drug as required by protocol
10. Be on stable antidiabetic treatment (insulin, oral agents, or lifestyle) that is not anticipated to change during the course of the study, except if medically required
11. Be on stable analgesic treatment (same medication and dose) or stable nonpharmacological pain treatment for at least 4 weeks prior to Screening (Visit 1) and remain on this stable treatment throughout the study (unless otherwise directed by a physician). Nonpharmacologic pain treatment includes the following: relaxation/hypnosis, physical or occupational therapy, counseling, etc. Episodic or periodic treatments such as monthly injections for treatment of pain (e.g., local anesthetics) will not be permitted.

EXCLUSION CRITERIA:

Patients with any one of the following will be excluded.

1. Patients with any condition that could interfere with the conduct of the study or confound efficacy evaluations including the following:

   1. Pain or neuropathy from another cause (including central pain, radiculopathy, painful arthritis, etc.)
   2. Skin or soft-tissue lesions in the area affected by neuropathy that are painful or could alter sensation
   3. Amputation, other than toes
2. Patients motivated by secondary gain, or where there is a negative-incentive to achieving pain and functional pain relief (eg, litigation). This will be determined by the patient's medical history.
3. Patients with clinically significant, progressive, or potentially unstable disease of any body system including cardiovascular, gastrointestinal, CNS, psychiatric, endocrine (other than diabetes), or immunologic, including patients with any of the following broad disease categories:

   1. Systemic infections (e.g., human immunodeficiency virus [HIV], hepatitis, tuberculosis [TB], syphilis)
   2. History of past (within the past 12 months) or present drug or alcohol abuse as per the Diagnostic and Statistical Manual - 4th Edition (DSM IV) criteria
   3. History of acute coronary syndrome within the past 12 months
   4. Active cancer within the previous 5 years
   5. Systemic chemotherapy or immunotherapy within the past 5 years
   6. History of major depression, bipolar disease, psychosis or suicidal ideation or attempts within the past 5 years
4. Patients with any of the following laboratory abnormalities at Screening (Visit 1) or Baseline (Visit 2):

   1. Clinically significant electrocardiogram (ECG) abnormality, including prolonged QTc (defined as QTc ≥ 450 msec)
   2. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 1.5 times the upper limit of normal (ULN)
   3. White blood cell (WBC) count ≤ 2500/μL, absolute neutrophil count ≤ 1000/μL, platelet count < 100,000
   4. Positive urine drug screen for drugs of abuse, except those prescribed by a properly licensed practitioner (e.g., opioids such as codeine for neuropathic pain)
   5. Other clinically significant laboratory values
5. Exposure to an investigational drug (including E2007) within the 30 days prior to Screening (Visit 1) or any prior exposure to E2007.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2007-06; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Laurenza, M.D., Study Director — Eisai Inc.
Locations (1):
- Dr. Richard Blonsky, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Perampanel 2mg: (Perampanel 2mg once daily for 15 weeks)
- Perampanel 4mg: (Perampanel 2mg once daily for 3 weeks, followed by perampanel 4mg once daily for 12 weeks)
- Perampanel 6mg: (Perampanel 2mg once daily for 3 weeks; followed by perampanel 4mg once daily for 3 weeks; and finally, perampanel 6mg once daily for 9 weeks)
- Perampanel 8mg: (Perampanel 2mg once daily for 3 weeks; then, perampanel 4mg once daily for 3 weeks; followed by perampanel 6mg once daily for 3 weeks; and finally, perampanel 8mg once daily for 6 weeks)
Period: Overall Study
Arm/Group | Placebo | Perampanel 2mg | Perampanel 4mg | Perampanel 6mg | Perampanel 8mg
Started | 73 | 72 | 69 | 68 | 70
Completed | 63 | 56 | 57 | 49 | 37
Not Completed | 10 | 16 | 12 | 19 | 33
Not completed — Adverse Event | 3 | 7 | 9 | 14 | 22
Not completed — Protocol Violation | 0 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 6 | 1 | 0 | 6
Not completed — Lack of Efficacy | 0 | 1 | 1 | 1 | 1
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0
Not completed — Other | 5 | 0 | 0 | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Perampanel 2mg | Perampanel 4mg | Perampanel 6mg | Perampanel 8mg | Total
Number analyzed (Participants) | 71 | 71 | 68 | 67 | 68 | 345
Age, Customized [Number; unit: Participants]
  <65 years | 50 | 50 | 40 | 34 | 41 | 215
  >=65 years | 21 | 21 | 28 | 33 | 27 | 130
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline characteristics look at Safety Population (subjects who were randomized, took at least 1 dose of study drug, and had at least 1 post-baseline assessment).
  Participants
    Female | 37 | 27 | 28 | 34 | 25 | 151
    Male | 34 | 44 | 40 | 33 | 43 | 194
Race/Ethnicity, Customized [Number; unit: participants] — This baseline characteristic is for Race.
  participants
    White | 56 | 56 | 56 | 60 | 60 | 288
    Black | 8 | 11 | 4 | 4 | 6 | 33
    Asian | 4 | 1 | 2 | 0 | 0 | 7
    Other | 3 | 3 | 6 | 3 | 2 | 17

OUTCOME MEASURES:

1. Primary Outcome: Change in Average Pain Scores From Baseline to Week 15/End of Treatment (EOT)
Description: Average of last 7 available scores prior to the visit, based on 11-point Likert-type numerical rating scale for pain (0=no pain, to 10=worst possible pain). This is based on a modified baseline observation carried forward (BOCF).
Time Frame: Baseline to Week 15/EOT
Population: Intent-to-Treat (ITT) Population - Randomized subjects who took at least 1 dose of study drug and had at least 1 efficacy assessment at Baseline.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo | Perampanel 2mg | Perampanel 4mg | Perampanel 6mg | Perampanel 8mg
Number analyzed (Participants) | 73 | 72 | 69 | 68 | 70
Scores on a Scale | -2.22 (2.19) | -1.73 (2.34) | -1.30 (2.18) | -1.85 (2.01) | -1.18 (2.00)

2. Primary Outcome: Responder Rate: Analysis of the Change in Pain Score From Baseline to Week 15/EOT in Subjects Who Had at Least a 30% Reduction in Pain Score
Description: Average pain scores were calculated as the average of last 7 available scores prior to the visit, based on 11-point Likert-type numerical rating scale for pain (0=no pain, to 10=worst possible pain). This is based on a modified BOCF.
Time Frame: Baseline to Week 15/EOT
Population: ITT Population. A responder was defined as a subject who had at least a 30% reduction in average pain scores from Baseline to Week 15/EOT.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Perampanel 2mg | Perampanel 4mg | Perampanel 6mg | Perampanel 8mg
Number analyzed (Participants) | 73 | 72 | 69 | 68 | 70
Percentage of Participants
  Responders (Yes) | 56.3 | 36.6 | 32.4 | 39.4 | 31.9
  Non-responders (No) | 43.7 | 63.4 | 67.6 | 60.6 | 68.1

3. Primary Outcome: Responder Rate: Analysis of the Change in Pain Score From Baseline to Week 15/EOT in Subjects Who Had at Least a 50% Reduction in Pain Score
Description: as for outcome 2
Time Frame: Baseline to Week 15/EOT
Population: ITT Population. A responder was defined as a subject who had at least a 50% reduction in average pain scores from Baseline to Week 15/EOT.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Perampanel 2mg | Perampanel 4mg | Perampanel 6mg | Perampanel 8mg
Number analyzed (Participants) | 73 | 72 | 69 | 68 | 70
Percentage of Participants
  Responders (Yes) | 38 | 23.9 | 22.1 | 30.3 | 18.8
  Non-responders (No) | 62 | 76.1 | 77.9 | 69.7 | 81.2

4. Primary Outcome: Mean Change in Average Pain Scores From Baseline at Each Study Week
Description: Average pain scores were calculated as the average of last 7 available scores prior to the visit, based on 11-point Likert-type numerical rating scale for pain (0=no pain, to 10=worst possible pain). Last on-treatment value refers to last 7 days of available diary data while subject was on double-blind study drug.
Time Frame: Baseline, Week 1 to Week 17
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo | Perampanel 2mg | Perampanel 4mg | Perampanel 6mg | Perampanel 8mg
Number analyzed (Participants) | 73 | 72 | 69 | 68 | 70
Scores on a Scale
  Week 1 | -0.58 (1.46) | -0.71 (1.33) | -0.58 (1.39) | -0.79 (1.44) | -0.72 (1.33)
  Week 2 | -0.87 (1.65) | -1.09 (1.53) | -0.80 (1.55) | -1.19 (1.71) | -1.05 (1.52)
  Week 3 | -1.19 (1.85) | -1.33 (1.64) | -0.91 (1.67) | -1.53 (1.92) | -1.22 (1.75)
  Week 4 | -1.46 (1.73) | -1.33 (2.01) | -1.10 (1.93) | -1.75 (1.99) | -1.38 (1.97)
  Week 5 | -1.49 (1.71) | -1.55 (2.21) | -1.12 (2.08) | -1.93 (1.96) | -1.56 (1.94)
  Week 6 | -1.73 (1.81) | -1.70 (2.17) | -1.31 (2.12) | -2.03 (2.14) | -1.58 (2.11)
  Week 7 | -1.99 (1.96) | -1.84 (2.10) | -1.50 (2.04) | -2.31 (2.32) | -1.80 (1.98)
  Week 8 | -1.91 (2.01) | -1.86 (2.05) | -1.72 (2.20) | -2.19 (2.23) | -1.71 (2.18)
  Week 9 | -2.19 (2.10) | -1.86 (2.14) | -1.76 (2.19) | -2.28 (2.12) | -2.01 (2.31)
  Week 10 | -2.30 (1.96) | -1.88 (2.19) | -1.84 (2.12) | -2.04 (1.98) | -1.92 (2.08)
  Week 11 | -2.39 (2.03) | -1.98 (2.20) | -1.85 (2.14) | -2.10 (2.09) | -1.95 (2.06)
  Week 12 | -2.46 (1.99) | -1.81 (2.31) | -1.76 (2.16) | -2.13 (2.11) | -1.91 (2.16)
  Week 13 | -2.36 (2.00) | -1.80 (2.16) | -1.62 (2.29) | -2.23 (1.99) | -2.01 (2.17)
  Week 14 | -2.30 (2.17) | -1.84 (2.31) | -1.56 (2.27) | -2.25 (2.00) | -1.89 (2.19)
  Week 15 | -2.39 (2.23) | -1.99 (2.39) | -1.58 (2.16) | -2.36 (1.91) | -1.93 (2.23)
  Week 16 | -2.40 (2.38) | -2.49 (2.20) | -1.50 (2.12) | -1.87 (2.12) | -1.88 (2.01)
  Week 17 | NA (NA) — Data unavailable for some arms due to end of study. | -5.50 (3.33) | NA (NA) — Data unavailable for some arms due to end of study. | NA (NA) — Data unavailable for some arms due to end of study. | 0.71 (NA) — Data unavailable for some arms due to end of study.
  Last On-Treatment Value | -2.24 (2.18) | -1.79 (2.32) | -1.48 (2.23) | -2.41 (2.15) | -1.69 (2.24)

5. Secondary Outcome: Change in Average Sleep Interference Scores From Baseline to Week 15/EOT
Description: Average of last 7 available scores prior to the visit, based on 11-point Likert-type numerical rating scale for sleep interference (0=pain did not interfere with sleep, to 10=pain completely interfered with sleep [unable to sleep]). Based on modified BOCF.
Time Frame: Baseline to Week 15/EOT
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo | Perampanel 2mg | Perampanel 4mg | Perampanel 6mg | Perampanel 8mg
Number analyzed (Participants) | 73 | 72 | 69 | 68 | 70
Scores on a Scale | -2.17 (2.18) | -1.49 (2.11) | -1.08 (2.19) | -1.71 (2.00) | -1.15 (2.19)

6. Secondary Outcome: Change in Short Form - McGill Pain Questionnaire (SF-MPQ) From Baseline to Week 15/EOT
Description: SF-MPQ sensory score = sum of intensity scores for descriptors 1-11 (throbbing, shooting, stabbing, sharp, cramping, gnawing, hot-burning, aching, heavy, tender, splitting). Each descriptor scored as 0=none, 1=mild, 2=moderate, or 3=severe. Range of possible sensory scores, 0 to 33, with a score of 33 being the most severe intensity.
Time Frame: Baseline and Week 15/EOT
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo | Perampanel 2mg | Perampanel 4mg | Perampanel 6mg | Perampanel 8mg
Number analyzed (Participants) | 73 | 72 | 69 | 68 | 70
Scores on a Scale | -5.6 (6.83) | -3.9 (6.93) | -4.8 (5.83) | -6.2 (6.91) | -2.9 (5.85)

7. Secondary Outcome: Analysis of Patient Global Impression of Change (PGIC) at Week 15/EOT
Description: At the EOT (Visit 7) or Early Withdrawal Visit (as appropriate), the subject assessed his/her status compared to how they felt before entering the study. This assessment included an evaluation of pain frequency and intensity, the occurrence of AEs, and overall functional status using a 7-point scale where 1=very much improved and 7=very much worse. Using Modified BOCF.
Time Frame: Week 15/EOT
Population: Subset of ITT population used, including subjects that completed PGIC at Week 15 visit, and using BOCF (baseline observation carried forward) subjects that terminated prior to Week 15 received a 'No Change' if due to AE or Lack of Therapeutic Efficacy, subjects who discontinued due to other reasons used PGIC scores from Early Termination visit.
Measure: Number; unit: Participants
Arm/Group | Placebo | Perampanel 2mg | Perampanel 4mg | Perampanel 6mg | Perampanel 8mg
Number analyzed (Participants) | 66 | 62 | 66 | 62 | 58
Participants
  Very much improved | 9 | 3 | 4 | 3 | 4
  Much improved | 17 | 13 | 15 | 14 | 8
  Minimally improved | 18 | 18 | 20 | 13 | 10
  No change | 18 | 24 | 24 | 28 | 31
  Minimally worse | 3 | 3 | 3 | 3 | 4
  Much worse | 1 | 1 | 0 | 1 | 1

8. Secondary Outcome: Change From Baseline to Week 15/EOT in SF-36 Physical and Mental Component Scores
Description: Short Form 36 Health Survey Questionnaire (SF-36) measuring limitations in Physical Components including physical activities, usual role activities (due to physical problems), measuring bodily pain, general health perceptions, and Mental Components including social activities, usual role activities (due to emotional problems), vitality (energy and fatigue. Each of the 8 domains are described by a score ranging from 0 to 100, for a range of total possible scores of 0-400 for physical and 0-400 for mental. Higher scores reflect better subject status.
Time Frame: Baseline and Week 15/EOT
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo | Perampanel 2mg | Perampanel 4mg | Perampanel 6mg | Perampanel 8mg
Number analyzed (Participants) | 73 | 72 | 69 | 68 | 70
Scores on a Scale
  Physical Component Score | 4.32 (7.43) | 1.57 (6.35) | 1.67 (8.21) | 1.59 (7.92) | 0.89 (6.86)
  Mental Component Score | -0.26 (9.14) | 0.40 (8.26) | 0.06 (10.77) | -1.90 (8.74) | -1.61 (9.56)

9. Secondary Outcome: Change From Baseline to Week 15/EOT in Hospital Anxiety and Depression Scale (HADS) Anxiety and Depression Subscale Scores
Description: HADS anxiety subscale score=sum of scores for 7 anxiety items, each scored on a 4-pt scale (0, 1, 2, or 3), where a higher score indicates worse anxiety. Range of possible HADS anxiety subscale scores, 0 to 21. HADS depression subscale score=sum of scores for 7 depression items, each scored on a 4-pt scale (0, 1, 2, or 3), where a higher score indicates worse depression. Range of possible HADS depression subscale scores, 0 to 21.
Time Frame: Baseline and Week 15/EOT
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo | Perampanel 2mg | Perampanel 4mg | Perampanel 6mg | Perampanel 8mg
Number analyzed (Participants) | 73 | 72 | 69 | 68 | 70
Scores on a Scale
  Anxiety | -0.5 (3.01) | -0.3 (2.85) | -0.5 (3.43) | -0.5 (2.89) | -0.4 (2.71)
  Depression | -0.7 (2.72) | -0.4 (2.43) | 0.0 (3.16) | 0.1 (3.42) | 0.2 (2.90)

10. Secondary Outcome: Withdrawal Due to Treatment Failure During Double-Blind Dosing Period
Description: Based on data reported on the End of Study case report form (CRF): If a subject terminated the study early during the Double-blind Dosing Period due to 'lack of therapeutic efficacy,' the subject was counted as a withdrawal due to treatment failure.
Time Frame: Baseline and Week 15
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Perampanel 2mg | Perampanel 4mg | Perampanel 6mg | Perampanel 8mg
Number analyzed (Participants) | 73 | 72 | 69 | 68 | 70
Participants
  Yes (withdrawn) | 0 | 1 | 1 | 1 | 1
  No (Not withdrawn) | 73 | 71 | 68 | 67 | 69

11. Secondary Outcome: Presence or Absence of Allodynia at Week 15/EOT
Description: Investigators rated subjects' allodynia as mild, moderate, severe, or not present. The presence of allodynia (yes/no) at Week 15/EOT was analyzed.
Time Frame: Week 15/EOT
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Perampanel 2mg | Perampanel 4mg | Perampanel 6mg | Perampanel 8mg
Number analyzed (Participants) | 73 | 72 | 69 | 68 | 70
Participants
  Yes (Allodynia present) | 20 | 18 | 19 | 17 | 17
  No (Allodynia absent) | 47 | 45 | 47 | 48 | 44

12. Secondary Outcome: Analysis of Rescue Analgesic Medication Use (Acetaminophen) During Double-Blind Dosing Period
Description: If acetaminophen was not reported on the Pain Therapy CRF or on the Concomitant Medication CRF, it was assumed that the subject did not use rescue analgesic medication.
Time Frame: Baseline to Week 15
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Perampanel 2mg | Perampanel 4mg | Perampanel 6mg | Perampanel 8mg
Number analyzed (Participants) | 73 | 72 | 69 | 68 | 70
Participants
  Yes (Used rescue analgesic medication) | 13 | 9 | 10 | 10 | 13
  No (Did not use rescue analgesic medication) | 60 | 63 | 59 | 58 | 57

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs): started on or after (or before if TEAE worsened in severity after first dose) the day of first dose of double-blind study drug up to 30 days after the last dose of double-blind study drug.
Arm/Group | Placebo | Perampanel 2mg | Perampanel 4mg | Perampanel 6mg | Perampanel 8mg
Serious Adverse Events (participants affected / at risk) | 2/71 | 2/71 | 2/68 | 8/67 | 8/68
Other Adverse Events (participants affected / at risk) | 26/71 | 30/71 | 33/68 | 40/67 | 38/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=71) | Perampanel 2mg (N=71) | Perampanel 4mg (N=68) | Perampanel 6mg (N=67) | Perampanel 8mg (N=68)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Cardiac Failure Congestive (Cardiac disorders) | 0 | 0 | 1 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Multi-organ Failure (General disorders) | 0 | 0 | 0 | 0 | 1
Death (General disorders) | 1 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0 | 2 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Escherichia Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Labyrinthitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Wound Infection Staphylococcal (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Blood Pressure Systolic Increased (Investigations) | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Balance Disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Homocidal Ideation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Suicide Attempt (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Renal Failure Acute (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1
Diabetic Neuropathy (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Urinary Retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Bronchial Hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Blood Pressure Fluctuation (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=71) | Perampanel 2mg (N=71) | Perampanel 4mg (N=68) | Perampanel 6mg (N=67) | Perampanel 8mg (N=68)
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 1 | 2 | 4
Nausea (Gastrointestinal disorders) | 2 | 4 | 2 | 5 | 5
Fatigue (General disorders) | 1 | 0 | 3 | 4 | 4
Gait Disturbance (General disorders) | 0 | 2 | 3 | 5 | 3
Oedema Peripheral (General disorders) | 5 | 3 | 5 | 3 | 2
Nasopharyngitis (Infections and infestations) | 3 | 2 | 5 | 1 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 5 | 3 | 2 | 3 | 4
Contusion (Injury, poisoning and procedural complications) | 3 | 1 | 3 | 4 | 5
Fall (Injury, poisoning and procedural complications) | 2 | 2 | 4 | 7 | 7
Blood Glucose Increased (Investigations) | 0 | 4 | 0 | 3 | 0
Weight Increased (Investigations) | 2 | 0 | 2 | 1 | 4
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 4 | 2 | 4 | 2
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 5 | 3 | 4 | 4
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 3 | 0 | 2 | 6 | 1
Dizziness (Nervous system disorders) | 1 | 6 | 2 | 15 | 15
Headaches (Nervous system disorders) | 5 | 2 | 3 | 3 | 4
Somnolence (Nervous system disorders) | 2 | 2 | 9 | 5 | 11
Insomnia (Psychiatric disorders) | 4 | 1 | 3 | 3 | 1
Hypertension (Vascular disorders) | 3 | 1 | 4 | 2 | 1
Orthostatic Hypotension (Vascular disorders) | 0 | 0 | 4 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No